CLINICAL TRIAL: NCT06608797
Title: Testing the Feasibility of Computer-based Cognitive Training in Individuals with Multiple Sclerosis Living in the Community
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Silvana Costa, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-1259-24
Record Dates: First submitted 2024-09-13; First posted 2024-09-23 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: learning, memory, cognitive training
MeSH Terms: conditions — Multiple Sclerosis | interventions — Educational Status; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training (Experimental): Computer based cognitive training delivered remotely via Zoom Health
  Interventions: Behavioral: Learning and memory training
- sham comparator (Sham Comparator): The sham comparator group will receive sham memory exercises administered on a laptop computer via Zoom Health twice a week for five weeks (10 placebo control sessions).
  Interventions: Behavioral: Sham Comparator

INTERVENTIONS:
Behavioral: Learning and memory training — The experimental group will receive memory retraining exercises administered on a laptop computer via Zoom Health twice a week for five weeks (10 training sessions).
  Arms: Training
Behavioral: Sham Comparator — The sham comparator group will receive sham memory exercises administered on a laptop computer via Zoom Health twice a week for five weeks (10 placebo control sessions).
  Arms: sham comparator

SUMMARY:
Cognitive impairments are common in multiple sclerosis (MS) diagnosed both at the onset and throughout the disease course. Poor cognitive abilities have been associated with poor outcomes such as higher levels of unemployment, poor quality of life, driving difficulties among others. Learning and memory are a common cognitive deficit. This computer-based cognitive training is a 10-session treatment proven to be effective in ameliorating learning and memory in individuals with MS across 3 realms of functioning: objective cognitive performance, daily life activities and neuroimaging. Despite this strong efficacy, as well as the recent clinical application of this computer-based cognitive training across the world, recent in-person studies have highlighted that transportation to the clinic to complete treatment sessions is a significant obstacle to clinical use of this effective treatment. To address this limitation, the proposed pilot study will test the efficacy of the computer-based cognitive training administered remotely via zoom health in persons with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* English as primary language
* Diagnosis of multiple sclerosis

Exclusion Criteria:

* Most recent exacerbation within one month
* Other Neurological History: head injury, stroke, seizures, or any other significant neurological history will not be included in the study
* Individuals with an active diagnosis of Major Depressive Disorder, Schizophrenia, Bipolar Disorder I or II will be excluded from the study.
* Poor Visual Acuity (corrected vision in worse eye < 20/60), diplopia, or nystagmus
* Inability to understand directions and following one, two, and three step commands
* Intact New Learning and Memory: Only individuals that show impaired performance on a memory test will be included in the study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
California Learning Verbal Test III | Primary outcome will be assessed at baseline (1 week before training start) and immediate follow-up (within 1 week after training completion)

SECONDARY OUTCOMES:
Ecological Memory Simulations | Secondary outcome will be assessed at baseline (1 week before training start) and immediate follow-up (within 1 week after training completion)

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
This is pilot data for potential future funding